CLINICAL TRIAL: NCT05358613
Title: Early Intervention Programs for at Risk Use of Psychoactive Substances and Gambling: ''My Choices'' Family
Brief Title: My Choices: Efficacy and Implementation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Joël Tremblay, Professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER-18-251-10.02
Record Dates: First submitted 2022-04-12; First posted 2022-05-03 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Alcohol Use Disorder, Mild; Alcohol Use, Unspecified
Keywords: Alcohol; Treatment
MeSH Terms: conditions — Alcoholism; Lymphoma, Follicular; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either receive the treatment now (10 working days, experimental group) or in 3 months (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (Experimental): The My Choices program will be offered immediately (maximum 10 working days from their first research interview) to the participants of this group.
  The treatment will be dispensed as usual, wich means there are no special conditions that need to be respected specifically for the study.
  Interventions: Behavioral: My Choices
- Waiting list (Active Comparator): The My Choices program will be offered 3 months after the first research interview to the participants in this group.
  The treatment will be dispensed as usual, wich means there are no special conditions that need to be respected specifically for the study.
  Interventions: Behavioral: My Choices

INTERVENTIONS:
Behavioral: My Choices — The My Choices program is an harm reduction program to modify substance use habits. It is based on the Miller & Rollnick Motivational interviewing as well as Deci and Ryan's Self-determination theory and Bandura's social learning theory.
  It is presented as a guide, divided in 6 phases. In every phase, participants will find, in the guide, some auto-observation exercises about their alcohol use habits and other aspects about their quality of life, reflexions and information about alcohol. The participants are also invited to note the number of standard units of alcohol they use on every occasion.
  Other Names: Alcochoix+

SUMMARY:
The aim of the study is to assess the efficacy of the My Choices - Alcohol program by comparing alcohol-use of people before and after doing the program to people that did not do the program on the same period of time (3 months).

DETAILED DESCRIPTION:
People with an alcohol addiction problem consume an average of 26.3 (sd = 12.4) drinks per week (Cournoyer et al., 2010). To observe a decrease of 25% in this average number of drinks for the group participating in the program " My Choices " immediately compared to the delayed group at 3 months, we need a sample size of 100 participants. This calculation assumes an alpha of 5%, a power of 80% and unbalanced groups due to the randomization method used. Considering an attrition rate of 11.3% at 3 months and 20% at 6 months (Tremblay et al., Submitted), it will be necessary to recruit at least 120 participants to maintain the required number for analyses.

References Cournoyer, L.-G., Simoneau, H., Landry, M., Tremblay, J., & Patenaude, C. (2010). Évaluation d'implantation du programme Alcochoix+ (FQRSC #2008-TO-120890). F. q. d. r. s. l. s. e. l. culture.

Tremblay, J., Dufour, M., Bertrand, K., Saint-Jacques, M., Ferland, F., Blanchette-Martin, N., Savard, A.-C., Côté, M., Berbiche, D., & Beaulieu, M. (Submitted). Efficacy of a Randomized Controlled Trial of Integrative Couple Treatment for Pathological Gambling (ICT-PG): 10-Month Follow-Up. Journal of Consulting and Clinical Psychology.

ELIGIBILITY:
Inclusion Criteria:

* Adults with at risk alcohol use (alcohol use over the Canadian low-risk alcohol drinking guidelines, without or with low consequences associated with their alcohol use).

Exclusion Criteria:

* Score at the DEBA (Assessment and Screening of Assistance needs) indicates a need for specialized treatment.
* Hospitalization for mental health problems in the last 30 days
* People with unstable mental health condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-05-14 (Actual)

PRIMARY OUTCOMES:
Change in self-reports of alcohol with the time-line follow-back (TLFB) in the last 90 days | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  The timeline follow-Back is a research tool to obtain self-reported quantitatives estimates of alcohol used every day in the last 3 months in term of standard drink. (Sobell & Sobell)
  Participants are asked in the first interview (2 weeks within eligibility evaluation) to remember day by day how many standard drinks they have had in the last 90 days.
Change in the Short Alcohol Dependance Data Questionnaire (SADD) | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  Short Alcohol Dependence Data questionnaire (SADD) is used to measure the severity of alcohol dependence. It comprises 15 items with a four-point frequency scale (never,sometimes, often, nearly always). A total score between 0 and 45 is obtained by adding the score from each of the items. Scores between 0 - 9 indicates low dependence, scores between 10 - 19 indicates medium dependence and a score of 20 or more indicates high dependence.
Change in the Inventory of consequences associated with alcohol use | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  It is a 7-items questionnaire, with a 0-10 (Never to always) scale that measures the consequences of alcohol consumption.
Change in the Severity of dependence scale (SDS) | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  The Severity of Dependence Scale (SDS) is a 5-item self-administered questionnaire that provides a score indicating the severity of dependence on drugs with a 4-point scale from 0 (Never) to 3 (Always). Score 0 indicates no dependence, score between 1-2 indicates low dependence, score between 3-5 indicates moderate dependance and score between 6 and 15 indicates a high dependance.

SECONDARY OUTCOMES:
Satisfaction with Life Domains Scale | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  20-items scale to assess the perceived quality of life. Participants can answer with 7 faces emojis (3 degrees of sadness, 3 degrees of happiness and 1 neutral).
Medical Outcomes Study-Social Support Survey (MOS-SSS) | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  8-items scale (Domains tangible and Emotional support), with a 5-point Likert scale ranging from 0 (None) to 4 (All of the time).
Readiness to change | 2 weeks within eligibility evaluation
  12-items scale with a 5 point Likert scale ranging from strongly disagree (-2) to strongly agree (2).
  This questionnaire assesses the motivation level to change alcohol use habits. The levels used are those of the transtheoretical model of change (Prochaska & DiClemente).
  The highest score indicates the stage in which the person is (precontemplation, contemplation or action) from a possibility from -8 to 8.
Motivations to change | 2 weeks within eligibility evaluation
  15-items scale with a 7 point Likert-like scale ranging from 1 (not at all) to 7 (Exactly) to assess the type of motivation that drives the person to modify his/her alcohol use habits.
  The questionnaire is based on the self-determination theory of Deci & Ryan.
  It is possible to assess the coefficient of self-determination by adding up the score of the identified and introjected motivation, and substracting to that score the external and amotivation scores. The higher is the coefficient of self-determination, the more internal is the motivation.
Generalized Anxiety Disorder (GAD-7) | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  Subjects are asked how often, during the last 2 weeks, they were bothered by each symptom. Response options were "not at all," "several days," "more than half the days," and "nearly every day," scored as 0, 1, 2, and 3, respectively (Löwe, Williams, Kroenke, Spitzer, 2006).
  A score between 0 and 4 means a minimal level of anxiety, between 5 and 9 means a mild level of anxiety, 10 to 14 means a moderate level of anxiety and a score between 15 and 21 means severe anxiety.
World Health Organization Well-Being Index (WHO-5) | 2 weeks within eligibility evaluation
  5-items scale with a 6 point Likert-like scale ranging from 0 (At no time) to 5 (All of the time). It is a subjective measure of the positive dimensions of mental health.
  Total score is between 0 to 100. Higher the score, better the level of well-being. A score under 50 could mean a higher risk of depression.
Impulsivity assessment with the Urgency, Premeditation (lack of), Perseverance (lack of), Sensation Seeking, Positive Urgency, Impulsive Behavior Scale, short version (UPPS-P short) | 2 weeks within eligibility evaluation
  It is a 20-items scale with a 4-point Likert-like scale from 1 (Agree strongly) to 4 (Disagree strongly).
  The items are representing 5 factors, which are negative and positive Urgency, sensation seeking, premedition (lack of) and perseverance (lack of).
  Scores are between 4 and 16 for each factor. The higher the score, the more impulsive is the person.
Attention disorder and hyperactivity disorder (ADHD) assesment | 2 weeks within eligibility evaluation
  6-items scale with a 5-point Likert-like scale from Never to Really often. If a person answers often or really often 4 times or more, it means that the person shows symptoms associated with ADHD.
Patient Health Questionnaire (PHQ-9) | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  9-items scale with a 4-point Likert-like scale from 0 (Not at all) to 3 (Nearly every day). The total score is obtained by adding up the answer to every 9 items, ranging from 0 to 27. The score indicates the level of depression severity: 0-4 indicates none or minimal severity, 5-9 indicates a mild severity, 10-14 indicates a moderate severity, 15-19 indicates a moderately severe depression and 20-27 indicates a severe depression.
Work and social adjustment scale (WSAS) | 2 weeks within eligibility evaluation
  5-items scale with a 9 point scale from 0 (Not at all) to 8 (very severely). The total score can be obtain by adding up the score of every items. A score above 20 suggests moderately severe or worse impairment. Scores between 10 and 20 are associated with significant functional impairment. Scores below 10 appear to be associated with subclinical populations.
Perceived Improvement Questionnaire | 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  23-items scale with a 4 point-scale from ''Worse than before'' to ''Much better than before''. The ratings allow the participants to judge to what degree their life has improved in 23 domains since the last 3 months.
Client Satisfaction Questionnaire (CSQ-3) | 3 months after first interview for the arm ''immediate treatment'' and 6 months after first interview for the group ''waiting list''
  3-items scale. The first item can be answered with a 4-point Likert-like scale from ''None of my needs were met'' to ''Almost all of my needs were met''. The second item can be answered with a 4-point Likert-like scale from ''Really satisfied'' to ''Really unsatisfied'' and the third item can be answered with a 4-point Likert-like scale from ''No, definitely not'' to ''Yes, definitely''.
Scale to Assess the Therapeutic Relationship-Client (STAR-C) | 3 months after first interview for the arm ''immediate treatment'' and 6 months after first interview for the group ''waiting list''
  12-items scale, with three domains (positive collaboration, emotional difficulties and positive clinician input), with a 5-point Likert-like scale ranging from 0 (Never) to 4 (Always).
  Total score can range from 0 to 48. The score can be obtained by adding up the score of every item. The scores from the ''emotional difficulties'' domain must be reversed. The higher the score the better is the therapeutic relationship.
Perception of reaching the goal | 3 months after first interview for the arm ''immediate treatment'' and 6 months after first interview for the group ''waiting list''
  Participants are asked to what extent they reached their goal about their alcohol use on a scale from 0 (Not at all) to 10 (Totally).
Difficulties associated with the alcohol-use | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  The participants are asked to what extent their alcohol use has caused them difficulties in the last 12 months, with a scale from 0 (Not at all) to 10 (Extremely).
Importance of change | 2 weeks within eligibility evaluation
  The participants are asked: to what extent is it important for you to change your alcohol use habits, with a scale from 0 (Not at all) to 10 (Extremely).
Perception of actual alcohol use | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  The participants are asked: what do you currently think about your alcohol-use? with a scale from 0 (Not at all) to 10 (Extremely).
Confidence to reach the alcohol use goal | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  The participants are asked: How confident are you of reaching your goals about your alcohol-use? with a scale from 0 (Not at all) to 10 (Extremely).
High-risk situations of alcohol use assessment | 2 weeks within eligibility evaluation, 3 and 6 months after first interview (The first admission has been October 28th and the last one is anticipated June 30th)
  Questionnaire to assess the situations in which the person is more at risk to drink and the level of confidence to not drink in this situation. The items are measured with a 0 (Never) to 10 (Always) Likert-like scale.

CONTACTS AND LOCATIONS:
Overall Officials: Joël Tremblay, Ph.D., Principal Investigator — Université du Québec à Trois-Rivières
Locations (5):
- Canada (5):
  - Centre Intégré Universitaire de Santé et de Services Sociaux du Saguenay-Lac-Saint-Jean, Jonquière, Quebec
  - Centre Intégré de Santé Services Sociaux de Laval, Laval, Quebec
  - Centre intégré de Santé et de Services Sociaux de Chaudière-Appalaches, Lévis, Quebec
  - Centre Intégré Universitaire de Santé et de Services Sociaux de la Capitale-Nationale, Québec
  - Université du Québec à Trois-Rivières, Québec

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT05358613/ICF_000.pdf